CLINICAL TRIAL: NCT05827510
Title: Fractional Radiofrequency for Treatment of Acne Scars and Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-585F_200
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Acne; Wrinkle
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: The subjects will be enrolled and assigned into two study groups, according to their indication; group A (acne scars) and B (facial wrinkles), each study group will receive treatment of different conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Acne scars (Experimental): All subjects will be treated with the BTL-585F system. Parameters' settings should be individually evaluated by the operator based on the treatment area and on the patient's medical and wound healing history. Parameters can be modified during subsequent visits, as per the practitioner's discretion.
  Interventions: Device: BTL-585F
- Facial wrinkles (Experimental): All subjects will be treated with the BTL-585F system. Parameters' settings should be individually evaluated by the operator based on the treatment area and on the patient's medical and wound healing history. Parameters can be modified during subsequent visits, as per the practitioner's discretion.
  Interventions: Device: BTL-585F

INTERVENTIONS:
Device: BTL-585F — BTL-585F device with BTL-585-4 applicator

SUMMARY:
This study will evaluate the clinical efficacy, safety and the performance of the fractional radiofrequency delivered by the BTL-585-4 applicator of the BTL-585F system for non-invasive treatment of acne scars and facial wrinkles. The study is a prospective multicenter open label two-arm study. The subjects will be enrolled and assigned into two study groups, according to their indication; group A (acne scars) and B (facial wrinkles), each study group will receive treatment of different conditions. Subjects of both groups will be required to complete three (3) treatment visits and two to three follow-up visits.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy, safety and the performance of the fractional radiofrequency delivered by the BTL-585-4 applicator of the BTL-585F system for non-invasive treatment of acne scars and facial wrinkles. The study is a prospective multicenter open label two-arm study. The subjects will be enrolled and assigned into two study groups, according to their indication; group A (acne scars) and B (facial wrinkles), each study group will receive treatment of different conditions. Subjects of both groups will be required to complete three (3) treatment visits and two to three follow-up visits.

At the baseline visit, health status will be assessed and, if needed, additional tests will be performed. Inclusion and exclusion criteria will be verified and informed consent will be signed. In addition photographs of the treated area will be taken.

The treatment administration phase in both study groups will consist of three (3) treatment visits, delivered 2-5 weeks apart. Subjects of both groups will receive treatment with the insulated or non-insulated microneedle tip (BTL-585-4-5 or BTL-585-4-6), depending on patients' skin sensitivity, followed by the application of superficial tip 32 (BTL-585-4-7) or 64 (BTL-585-4-8), depending on the size of the treatment site. Treatment settings will be adjusted individually according to the severity of the subjects' condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment and reduction of facial wrinkles or acne scars
* Subjects should be able to understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible wrinkles or acne scars in the treated area when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 6 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* History of skin disorders, keloids, very dry and fragile skin
* Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks
* Botox®/collagen/fat injections or other injected bio-material in the treated area within three months prior to the treatment
* Use of non-steroidal anti-inflammatory drugs one week before and after each treatment session
* Treating over tattoo or permanent make-up
* Treating over eyelids or the lips
* Patients with allergy to anesthetics should not be treated under anesthesia
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use ani-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* Any other disease or condition (e.g. eye disease) at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Change in wrinkle severity | 5 months
  Evaluation of wrinkle severity based on photographs before and after the study procedure.
Change in acne scars | 5 months
  Evaluation of improvement in acne scars based on photographs before and after the study procedure.

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events [Safety and Tolerability] | 5 months
  Evaluation of the safety of the BTL-585F device with BTL-585-4 applicator for non-invasive reduction of wrinkles and treatment of acne scars by monitoring of adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Precision Skin Institute, Davie, Florida
  - Yael Halaas, M.D., FACS, New York, New York

IPD SHARING:
Plan to Share IPD: No